CLINICAL TRIAL: NCT04713982
Title: Impact of Deutetrabenazine on Functional Speech and Gait Dynamics in Huntington Disease
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, Amy E Brown, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200069
Record Dates: First submitted 2021-01-06; First posted 2021-01-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — deutetrabenazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Deutetrabenazine (Experimental): The mode of administration is oral. Subjects will be started on deutetrabenazine at a dose of 6mg/day. Dosing will be up-titrated in increments of 6mg/day per week to achieve optimal chorea control.
  Interventions: Drug: Deutetrabenazine

INTERVENTIONS:
Drug: Deutetrabenazine — Maximum dose of 48mg/day or up to 36 mg/d if receiving a strong CYP2D6 inhibitor
  Other Names: Austedo

SUMMARY:
Examine the effects of deutetrabenazine on functional speech and gait impairment

DETAILED DESCRIPTION:
This is a two-year, prospective, single-arm study examining the effects of deutetrabenazine on functional speech and gait impairment. Participants will undergo comprehensive evaluations of speech production, fine motor skills, gait, and balance both before and after the initiation of deutetrabenazine. The investigators will utilize a variety of standardized, well-validated assessments as well as 3D motion analysis of both speech and gait parameters to determine the functional impact of deutetrabenazine on speech and motor performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HD with documented CAG repeat ≥ 37
* UHDRS total maximal chorea score of ≥ 8
* Able to walk at least 10 meters
* Medically stable outpatient, based on the investigator's judgment
* Willing and able to give written informed consent prior to performing any study procedures
* Have completed at least 10th grade
* Montreal Cognitive Assessment score ≥ 22 on screening
* Female subjects of childbearing potential agree to use an acceptable method of contraception from screening through study completion

Exclusion Criteria:

* Severe depression or suicidal ideation
* History of suicidal behavior
* Unstable or serious medical or psychiatric illness
* Renal or hepatic impairment
* Severe speech impairment or anarthria
* Inability to swallow study medication
* Women who are pregnant or breast feeding
* History of alcohol or substance abuse within the last 12 months
* Current use of VMAT2 inhibitor (tetrabenazine, deutetrabenazine, valbenazine)
* Concurrent participation in any other investigational drug trials
* EKG QTcF> 500 mse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Sentence Intelligibility Test (SIT) | Up to 10 weeks
  SIT is a measure of speech intelligibility that requires the participant to read aloud 11 sentences that increase in length from 5 to 10 words. Speech intelligibility is indexed in terms of percent intelligible. This is determined by calculating the mean number of correct words transcribed from the SIT transcriptions by three unfamiliar listeners and dividing this by the total number of words in the 11-sentence sample.
Motor Speech Evaluation (MSE) | Up to 10 weeks
  The MSE will include a set of tasks described by Duffy (2013) that permit consistent rating of perceptual characteristics associated with motor speech disorders. These tasks include vowel prolongation, alternating motion rates, sequential motion rates, and contextual speech (oral reading, picture description, conversational speech). These recordings will be used to complete the perceptual assessment of speech characteristics using the Mayo Clinic classification system.

SECONDARY OUTCOMES:
3-D optical motion capture system recording | Up to 10 weeks
  To determine the effect of deutetrabenazine on facial movements at rest and during functional task performance (e.g., speaking, chewing) in individuals with HD, the investigators will utilize a 3-D optical motion capture system (Motion Analysis, Ltd.) consisting of six infrared Kestrel cameras with a sensor resolution of 2.2 million pixels at 2,048 x 1,088 full resolution. Facial movements will be captured by placing small (2mm) reflective spheres on each patient's jaw (right/left/center), mouth (right/left corner, upper/lower lip center), and cheeks (right/left zygomatic bone). Further, reflective markers will be placed on the forehead (right/left eyebrows, right/left forehead). Four head markers will serve as reference markers for head movement correction and transposition of all marker movement into a head-based coordinate system.
Functional Joint Kinematics Improvements | Up to 10 weeks
  To determine the effect of deutetrabenazine on joint kinematics and spatiotemporal parameters using 3D motion analysis. Participants will be recording using the Xsens MVN Awinda motion capture system during a 10 meter walk test. Lower- and upper-limb kinematics will be recorded. Wireless sensors will be placed on the ankle, thigh, hand, forearm, bicep, and head. The velocity of the 10 meter walk can be compared to age and gender matched normative values. Gait speed correlates with functional ability, balance and confidence. Three trials are completed, and the average of the three scores is documented. This test will be completed using the 3D motion analysis system.
Four Square Step Test (FSST) | Up to 10 Weeks
  The FSST assesses dynamic balance stepping over objects forward, backwards, and sideways. The individual is required to step as fast as possible into each square, requiring the individual to step objects in varying directions. Two tests are completed, with the best time documented as the score.
Functional Gait Assessment (FGA) | Up to 10 weeks
  The FGA assesses dynamic balance during gait and provides objective information regarding risk of falling. The FGA consists of ten items scored from 0-3, with a maximum total score of 30 points. Items include normal walking, walking with speed changes, walking with head turns, pivot turns, obstacle negotiation, tandem walking, walking with eyes closed, walking backward, and negotiating stairs. Scores less than 23/30 are predictive of falls.

OTHER OUTCOMES:
Communication Effectiveness Survey | Up to 10 weeks
  The CES is an 8-item patient reported outcome measure that is designed to rate communication effectiveness in individuals with dysarthria. Each of the items presents a communication situation (e.g., talking on the phone with a familiar listener; talking while driving in a car, etc.) and the participant rates his or her perceived ability to communicate in that situation on a scale from "1" (not at all effective) to "4" (very effective).
Nine-Hole Peg Test | Up to 10 weeks
  The Nine-Hole Peg Test is an assessment of fine motor coordination that measures each hand individually. The final score reported is the time required to place and remove nine pegs with each hand. Results are compared to age and gender matched normative values. This test will assess the impact of chorea on fine motor movements and dexterity.
10 Meter Walk test | Up to 10 Weeks
  With the 10 Meter Walk Test, velocity can be compared to age and gender matched normative values. Gait speed correlates with functional ability, balance and confidence. Three trials are completed, and the average of the three scores is documented. This test will be completed using the 3D motion analysis system.
Health Status | Up to 10 weeks
  The investigators will be using the short-form 36 (SF-36) which is a generic patient-reported outcome measure that quantifies perceived health status. It is used as a measure of health-related quality of life. Sub sections include physical function, role limitations secondary to physical problems, general health perceptions, vitality, social functioning, role limitations due to emotional problems, mental health, and health transition. Participants respond referring to their perceived health over the past 4 weeks.
The Functional Assessment of Chronic Illness Therapy (FACIT) scale | Up to 10 weeks
  The FACIT scale has been validated in a number of chronic conditions, including cancer, Parkinson's disease, multiple sclerosis, and HIV/AIDS (Webster 2003). It includes assessments of physical, social, emotional, and functional well-being and is available in multiple condition- and treatment-specific versions. The FACIT scale is sensitive to changes in individual participants over time and can also be used to compare patient populations.

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No